CLINICAL TRIAL: NCT04923516
Title: Prevalence of Acute Hepatic Porphyria in Population With Suggestive Clinical Picture
Brief Title: Prevalence of Acute Hepatic Porphyria
Acronym: PHA
Status: Completed | Type: Observational
Sponsor: Association pour la Recherche en Medecine Interne (Network)
Responsible Party: Sponsor
Other Study IDs: 2021-A00566-35
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Acute Hepatic Porphyria
MeSH Terms: conditions — Coproporphyria, Hereditary | interventions — Porphobilinogen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dosage of Delta-aminolevulinic acid and Porphobilinogen — Results of dosages of Delta-aminolevulinic acid and Porphobilinogen which are performed in accordance with the current practice will be recorded

SUMMARY:
To determine the proportion of patients suffering from acute hepatic porphyria (AHP) from different hospital departments and referred to an internist referent for a suggestive clinical picture with a first negative etiological assessment.

DETAILED DESCRIPTION:
In this context, this study aims to assess the prevalence of PHA in a population of patients with a suggestive clinical picture. A better knowledge of the pathology will make it possible to better guide patients and prevent them from diagnostic wandering fraught with physical and psychological consequences.

This is an observational, ambispective, transversal, multicenter study carried out in France. The goal is to recruit a cohort that will reflect current practice. 500 patients will be recruted.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 to 60;
* Presenting severe abdominal pain, afebrile and diffuse over several days, evolving for less than 5 years;
* With at least one of the following symptoms:

  * Peripheral neurological symptoms: decreased driving force and pain in the limbs (roots of the thighs), etc. ;
  * Central neurological symptoms: psychiatric (depression, anxiety, insomnia), disturbances of consciousness, etc. ;
  * Autonomous neurological symptoms: tachycardia, nausea, vomiting, constipation, etc.
* With a first negative etiological assessment requested by an emergency physician, gastroenterologist, gynecologist, neurologist, internist or another specialty, or with a diagnosis of acute hepatic porphyria less than 6 months;
* Patient able to understand the information related to the study and having indicated his non-objection to the collection of data concerning him;

Exclusion Criteria:

* Patient with a diagnosis of acute hepatic porphyria for more than 6 months;
* Patient unfit to participate in the study, due to cognitive or linguistic difficulties;
* Protected patient (under legal protection, or deprived of liberty by judicial or administrative decision).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The target population is made up of patients presenting signs suggestive of acute hepatic porphyria or recently diagnosed, from consultations with gastroenterologists, emergency physicians, neurologists, gynecologists, internists or other specialties, referred to an acute hepatic porphyria referent internist participating in the study, within the framework of of the etiological exploration of their clinical picture.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Binary criterion corresponding to the diagnosis of acute hepatic porphyria (acute hepatic porphyria + / acute hepatic porphyria -) via physiological parameter. | 1 day
  The diagnosis of acute hepatic porphyria is based on urine testing of the neurotoxic precursors of haem: Delta-aminolevulinic acid and Porphobilinogen. A patient will be considered to have acute hepatic porphyria (acute hepatic porphyria +) if:
  * Delta-aminolevulinic acid ≥ 3 µmol / mol Cr And or
  * Porphobilinogen ≥ 1 µmol / mol Cr Otherwise, the patient will be considered to be acute hepatic porphyria free (acute hepatic porphyria -).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No